CLINICAL TRIAL: NCT03796052
Title: A Single Center, Clinical Study to Determine the Safety and Efficacy of an Avena Sativa Skincare Regimen for Therapy-Related Pruritus and Xerosis in Cancer Patients
Brief Title: Study Determining Safety and Efficacy of Avena Sativa (Oat) Skincare Products for Treating Skin Dryness and Itching in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCSSKA000844
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Ichthyosis; Pruritus
Keywords: Pruritis; Itching; Dryness; Xerosis
MeSH Terms: conditions — Ichthyosis; Pruritus

STUDY DESIGN:
Intervention Model Description: All participants will receive the same study regimen consisting of 3 products: a body wash, a body cream, and an anti-itch balm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avena Sativa Skincare Regimen (Experimental): Avena sativa-containing body wash, body cream, and anti-itch balm
  Interventions: Other: Avena Sativa Skincare Regimen

INTERVENTIONS:
Other: Avena Sativa Skincare Regimen — Regimen consisting of 3 topical agents containing Avena Sativa (oat) kernel flour: a body wash (type = cosmetic), a body cream (type = cosmetic), and an anti-itch balm (type = OTC monograph drug with 0.5% Pramoxine HCl)

SUMMARY:
This study will test the safety and efficacy of three topical agents containing oat kernel flour to determine how well they relieve skin dryness and itching related to cancer therapies. Participants will receive a body wash, a body cream, and an anti-itch balm to use at home for 4-6 weeks.

DETAILED DESCRIPTION:
Many patients undergoing cancer therapies experience skin reactions like dry skin, rash, redness, itchiness, and hyperpigmentation. Dry skin and itching are especially common for those undergoing chemotherapy and targeted treatments.

Skincare products containing Avena sativa (oat) kernel flour have a long history of tolerance and efficacy in treating various skin conditions involving pruritus (itching) and xerosis (dry skin), as Avena sativa (oat) kernel flour is known for its skin protectant properties and soothing effects on skin. This study will evaluate the safety and efficacy of a regimen of three topical agents containing Avena sativa (oat) kernel flour for cancer patients experiencing mild to moderate pruritus and/or xerosis.

Participants will received the products at Baseline (Visit 1) and return to the clinical site at Week 5 +/- 1 week for Visit 2. In addition, questionnaires will be completed remotely between Baseline and Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* able to read, write, speak, and understand English
* has signed Informed Consent including Photograph Release
* has a prior diagnosis of a solid or hematologic tumor and either:

  1. is currently undergoing therapy with a systemic agent and has completed at least 3 cycles without severe skin reactions.
  2. has received therapy with a systemic agent in the past 28 days.
  3. is greater than 1 year status post allogeneic hematopoietic stem cell transplantation.
* is undergoing one or more types of cancer treatment that are commonly known to cause mild to moderate skin reactions such as rash, dryness, and/or itching
* is diagnosed with mild to moderate skin dryness (xerosis) and/or itching (pruritus).
* is capable of all self-care and is up and mobile at least 50% of the day
* intends to complete the study and is willing/able to follow all study instructions.

Exclusion Criteria:

* has known allergies or sensitivity to skincare products or study product ingredients.
* has other skin conditions or diseases that the investigator thinks would interfere with the study or put the subject at higher risk (e.g. immunosuppressive diseases, skin infections, etc.)
* has severe skin dryness, itching, or rash.
* is undergoing radiation therapy.
* is undergoing chemotherapy or adjuntive therapies known to commonly cause complex or severe skin reactions.
* has uncontrolled diabetes.
* is pregnant or planning to become pregnant during the study.
* is participating in another study for which the participant is receiving a treatment or therapy (observational studies are okay).
* is an employee or family member of the investigator, study site, or Sponsor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline to Visit 2 in CTCAE Grading of Xerosis | Baseline to Week 5 +/- 1 week
  The investigator will evaluate subjects for overall xerosis (skin dryness) using the Common Terminology Criteria for Adverse Events (CTCAE) grading scale. For xerosis, the scale ranges from 1 (dryness covering less 10% of body surface area and no associated erythema or pruritus) to 3 (dryness covering greater than 30% of body surface area and associated with itching; limits daily self care activities of daily living). A "0" grade will be used to document subjects with no presence of the CTCAE skin adverse event symptoms for xerosis. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in CTCAE Grading of Pruritus | Baseline to Week 5 +/- 1 week
  The investigator will evaluate subjects for overall pruritus (skin itching) using the Common Terminology Criteria for Adverse Events (CTCAE) grading scale. For pruritus, the scale ranges from 1 (Mild or localized; topical intervention indicated) to 3 (widespread and constant itching; limits daily self-care activities or sleep). A "0" grade will be used to document subjects with no presence of the CTCAE skin adverse event symptoms for pruritus. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Overall Xerosis Grading | Baseline to Week 5 +/- 1 week
  The investigator will evaluate subjects for overall xerosis (skin dryness) using a 0 (none) to 3 (severe) scale. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Overall Pruritus Grading | Baseline to Week 5 +/- 1 week
  The investigator will question subjects for overall pruritus (skin itching) using a 0 (none) to 3 (severe) scale. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Overall Irritation Assessment | Baseline to Week 5 +/- 1 week
  The investigator will evaluate subjects for overall irritation using a 0 (none) to 4 (very severe) scale. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).

SECONDARY OUTCOMES:
Frequency Distribution for Overall Tolerance at Visit 2 - Subject Rating | Week 5 +/- 1 week
  The subject will rate how well he/she tolerated the study regimen using the following choices: Well tolerated, tolerated, or not tolerated.
Frequency Distribution for Overall Tolerance at Visit 2 - Investigator Rating | Week 5 +/- 1 week
  The investigator will rate how well the participant tolerated the study regimen using the following choices: Well tolerated, tolerated, or not tolerated.
Mean Change from Baseline to Visit 2 in PRO-CTCAE Skin Dryness | Baseline to Week 5 +/- 1 week
  The Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) will be completed for Skin Dryness. The question asks subjects to rate the severity of their dry skin at its worst over the last 7 days from None to Very Severe on a 5-point scale. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in PRO-CTCAE Itching | Baseline to Week 5 +/- 1 week
  The Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) will be completed for Itching. The question asks subjects to rate the severity of their itchy skin at its worst over the last 7 days from None to Very Severe on a 5-point scale. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Skindex-16 Global Score | Baseline to Week 5 +/- 1 week
  The Skindex-16 is a dermatology-specific quality of life measuring tool. (The SKINDEX contact information and permission to use: Mapi Research Trust, Lyon, France. Internet: https://eprovide.mapi-trust.org). It contains 16 questions that ask subjects to rate how often over the last 7 days they have been bothered by various skin conditions on a scale of 0 (never bothered) to 6 (always bothered). The global score is the average score for all questions and is transformed to a linear scale ranging from 0 (never bothered) to 100 (always bothered) so a higher score indicates a lower quality of life. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Skindex-16 Emotional Subscale | Baseline to Week 5 +/- 1 week
  The Skindex-16 is a dermatology-specific quality of life measuring tool (The SKINDEX contact information and permission to use: Mapi Research Trust, Lyon, France. Internet: https://eprovide.mapi-trust.org). It contains 16 questions that ask subjects to rate how often over the last 7 days have they been bothered by various skin conditions on a scale of 0 (never bothered) to 6 (always bothered). The Emotional subscale looks at the average score of questions 5-11 regarding emotion; the emotional score is transformed to a linear scale ranging from 0 (never bothered) to 100 (always bothered) so a higher score indicates a lower quality of life. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Skindex-16 Symptoms Subscale | Baseline to Week 5 +/- 1 week
  The Skindex-16 is a dermatology-specific quality of life measuring tool (The SKINDEX contact information and permission to use: Mapi Research Trust, Lyon, France. Internet: https://eprovide.mapi-trust.org). It contains 16 questions that ask subjects to rate how often over the last 7 days have they been bothered by various skin conditions on a scale of 0 (never bothered) to 6 (always bothered). The Symptoms subscale looks at the average score of questions 1-4 individual responses regarding symptoms; the symptoms score is transformed to a linear scale ranging from 0 (never bothered) to 100 (always bothered) so a higher score indicates a lower quality of life. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Skindex-16 Functional Subscale | Baseline to Week 5 +/- 1 week
  The Skindex-16 is a dermatology-specific quality of life measuring tool (The SKINDEX contact information and permission to use: Mapi Research Trust, Lyon, France. Internet: https://eprovide.mapi-trust.org). It contains 16 questions that ask subjects to rate how often over the last 7 days have they been bothered by various skin conditions on a scale of 0 (never bothered) to 6 (always bothered). The Functional subscale looks at the average score of questions 12 - 16 regarding daily functioning; the functional score is transformed to a linear scale ranging from 0 (never bothered) to 100 (always bothered) so a higher score indicates a lower quality of life. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Skin Moisture | Baseline to Week 5 +/- 1 week
  Skin moisture will be measured with a Corneometer, with values ranging from 0 (no moisture) to 120 (most moisturized) arbitrary units. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Skin Water Loss | Baseline to Week 5 +/- 1 week
  The amount of water lost through the skin will be measured with a Vapometer. Higher numbers indicate more water loss. Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Self-Assessment of Dryness | Baseline to Week 5 +/- 1 week
  Subjects will be asked to rate their overall skin dryness on a scale of 1 (very dry) to 10 (skin feels moisturized). Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Self-Assessment of Flakiness | Baseline to Week 5 +/- 1 week
  Subjects will be asked to rate their overall skin flakiness on a scale of 1 (flaking very apparent) to 10 (no visible flaking). Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Self-Assessment of Itchiness | Baseline to Week 5 +/- 1 week
  Subjects will be asked to rate their overall skin itchiness on a scale of 1 (very itchy) to 10 (not at all itchy). Baseline will be compared to the subjects' final visit (Week 5 +/- 1 weeks).
Mean Change from Baseline to Visit 2 in Self-Assessment of Roughness | Baseline to Week 5 +/- 1 week
  Subjects will be asked to rate their overall skin roughness/texture on a scale of 1 (very rough) to 10 (not at all rough). Baseline will be compared to the subjects' final visit (Week 5 +/- 1 weeks).
Mean Change from Baseline to Visit 2 in Self-Assessment of Smoothness | Baseline to Week 5 +/- 1 week
  Subjects will be asked to rate their overall skin smoothness on a scale of 1 (not at all smooth) to 10 (very smooth). Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Self-Assessment of Softness | Baseline to Week 5 +/- 1 week
  Subjects will be asked to rate their overall skin softness on a scale of 1 (not at all soft) to 10 (very soft). Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Self-Assessment of Comfort | Baseline to Week 5 +/- 1 week
  Subjects will be asked to rate their overall skin comfort on a scale of 1 (uncomfortable/irritated) to 10 (very comfortable/not at all irritated). Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).
Mean Change from Baseline to Visit 2 in Self-Assessment of Overall Look/Feel | Baseline to Week 5 +/- 1 week
  Subjects will be asked to rate the overall look and feel of their skin on a scale of 1 (not healthy looking) to 10 (healthy looking). Baseline will be compared to the subjects' final visit (Week 5 +/- 1 week).

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lacouture, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.

REFERENCES:
- [Background] Kurtz ES, Wallo W. Colloidal oatmeal: history, chemistry and clinical properties. J Drugs Dermatol. 2007 Feb;6(2):167-70. PMID 17373175
- [Background] Fowler JF Jr. Colloidal oatmeal formulations and the treatment of atopic dermatitis. J Drugs Dermatol. 2014 Oct;13(10):1180-3; quiz 1184-5. PMID 25607551
- [Background] Ilnytska O, Kaur S, Chon S, Reynertson KA, Nebus J, Garay M, Mahmood K, Southall MD. Colloidal Oatmeal <em>(Avena Sativa)</em> Improves Skin Barrier Through Multi-Therapy Activity. J Drugs Dermatol. 2016 Jun 1;15(6):684-90. PMID 27272074
- [Background] Sur R, Nigam A, Grote D, Liebel F, Southall MD. Avenanthramides, polyphenols from oats, exhibit anti-inflammatory and anti-itch activity. Arch Dermatol Res. 2008 Nov;300(10):569-74. doi: 10.1007/s00403-008-0858-x. Epub 2008 May 7. PMID 18461339
- [Background] Criquet M, Roure R, Dayan L, Nollent V, Bertin C. Safety and efficacy of personal care products containing colloidal oatmeal. Clin Cosmet Investig Dermatol. 2012;5:183-93. doi: 10.2147/CCID.S31375. Epub 2012 Nov 8. PMID 23204849
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Elman S, Hynan LS, Gabriel V, Mayo MJ. The 5-D itch scale: a new measure of pruritus. Br J Dermatol. 2010 Mar;162(3):587-93. doi: 10.1111/j.1365-2133.2009.09586.x. Epub 2009 Dec 1. PMID 19995367
- [Background] Chren MM, Lasek RJ, Sahay AP, Sands LP. Measurement properties of Skindex-16: a brief quality-of-life measure for patients with skin diseases. J Cutan Med Surg. 2001 Mar-Apr;5(2):105-10. doi: 10.1007/BF02737863. Epub 2001 Mar 21. PMID 11443481
- [Background] Common Terminology Criteria for Adverse Events (CTCAE). (2018, Mar 01). Retrieved from https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm
- [Background] The PRO-CTCAE Measurement System. (2018, Sep 14). Retrieved from https://healthcaredelivery.cancer.gov/pro-ctcae/measurement.html
- [Background] Blume-Peytavi U, Kottner J, Sterry W, Hodin MW, Griffiths TW, Watson RE, Hay RJ, Griffiths CE. Age-Associated Skin Conditions and Diseases: Current Perspectives and Future Options. Gerontologist. 2016 Apr;56 Suppl 2:S230-42. doi: 10.1093/geront/gnw003. PMID 26994263
- [Background] Skin Conditions. (2012, Jun 26). Retrieved from https://www.cancer.net/navigating-cancer-care/side-effects/skin-conditions
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSSKA000844&attachmentIdentifier=48eeefb6-abfc-4be4-87ec-7d1620ff69d8&fileName=CCSSKA000844_Ribbons_Clinical_Study_Report_Synopsis_14OCT2020.pdf&versionIdentifier=